CLINICAL TRIAL: NCT01744782
Title: An Open-Label, Safety and Effectiveness Study of Cysteamine Bitartrate Delayed-release Capsules (RP103) in Cysteamine Treatment Naïve Patients With Cystinosis
Brief Title: Safety/Effectiveness Study of Cysteamine Bitartrate Delayed-release Capsules (RP103) in Cysteamine Treatment Naive Patients With Cystinosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP103-08
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cystinosis
Keywords: Nephropathic Cystinosis; Cysteamine; Delayed-release Cysteamine; CTNS Protein, Human; Orphan Disease
MeSH Terms: conditions — Cystinosis; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP103 (Experimental): From Day 1 and throughout the duration of participation, RP103 (Cysteamine Bitartrate Delayed-release Capsules) was administered every 12 hours (Q12H), supplied as 75 mg and 25 mg capsules.
  Interventions: Drug: RP103

INTERVENTIONS:
Drug: RP103 — Cysteamine Bitartrate Delayed-release Capsules (RP103) were administered twice daily, orally or via gastrostomy tube (G-tube), after a 2-hour fast. The starting dose was one-quarter of the RP103 targeted maintenance dose based on age, weight, and body surface area. The recommended targeted maintenance dose for children up to 6 years old was 1 gram/m²/day, in 2 divided doses given Q12H. The dose was gradually escalated, in 10% steps, based on monitoring of WBC cystine levels 30 minutes after the morning RP103 dose collected every 2 weeks, until the participant's WBC cystine level was <1 nmol ½ cystine/mg protein.
  Other Names: Cysteamine Delayed-release Capsules

SUMMARY:
This was a long-term, open-label study of the safety, tolerability and effectiveness of RP103 in cystinosis patients who were naïve to any form of cysteamine treatment. Participants received RP103 treatment for at least 12 months. U.S. participants transitioned to the commercially approved drug PROCYSBI®. In Brazil, after at least 12 months of study participation and upon approval by the Brazilian regulatory authorities, participants were eligible to transition to a post-study drug supply program, and continue to receive the drug at no personal cost.

DETAILED DESCRIPTION:
The purpose of this study was to gather information about the safety and effectiveness (how well it works to treat cystinosis) of a new drug called RP103.

In cystinosis, the body builds up cystine. When taken regularly, the active ingredient of an older, already approved drug called Cystagon® (cysteamine bitartrate) reduces cystine in the body. RP103 has the same active ingredient as Cystagon® and is designed to reduce cystine in a similar way that Cystagon® does. RP103 is also different from Cystagon®: Instead of the cysteamine bitartrate being absorbed from the stomach, RP103 is designed to be absorbed from the small intestine. This may make the effects of the drug last longer, so that it can be taken twice a day instead of four times a day like Cystagon®.

To decide if RP103 is effective, the study used two types of blood tests. One test is pharmacodynamics (PD), which measures the amount of white blood cell (WBC) cystine after taking study drug. WBC cystine is a laboratory test used to find out if cysteamine bitartrate is reducing cystine levels in the body. The second test is pharmacokinetics (PK), which measures the amount of cysteamine in the blood after taking the drug.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with a documented diagnosis of cystinosis
* No clinically significant change in liver function tests, i.e. 1.5 times upper limit of normal (ULN) for alanine aminotransferase (ALT) and aspartate aminotransferase (AST), and/or 1.5 times ULN for total bilirubin, within 6 months prior to Screening
* No clinically significant change in renal function, i.e. estimated glomerular filtration rate (GFR) within 6 months prior to Screening
* Must have an estimated GFR > 20 mL/minute/1.73m² (using the equation from Schwartz 2009 J Am Soc Nephrol 20:629-647)
* Female participants who are sexually active and of childbearing potential, i.e. not surgically sterile (tubal ligation, bilateral oophorectomy, or hysterectomy) or at least 2 years naturally postmenopausal must agree to use an acceptable form of contraception from Screening through completion of the study. Acceptable forms of contraception for this study include hormonal contraceptives (oral, implant, transdermal patch, or injection) at a stable dose for at least 3 months prior to Screening, barrier (spermicidal condom or diaphragm with spermicide), IUD, or a partner who has been vasectomized for at least 6 months. Childbearing potential was defined as a female who had reached menarche.
* Participant or their parent or guardian must provide written informed consent and assent (where applicable) prior to participation in the study
* Had not taken any form of cysteamine bitartrate in the past

Exclusion Criteria:

* Current history of the following conditions or any other health issues that make it, in the opinion of the Investigator, unsafe for study participation:
* Inflammatory bowel disease if currently active, or prior resection of the small intestine
* Heart disease (e.g., myocardial infarction, heart failure, unstable arrhythmias, or poorly controlled hypertension) within 90 days prior to Screening
* Active bleeding disorder within 90 days prior to Screening
* History of malignant disease within 2 years prior to Screening
* Hemoglobin level of < 10 g/dL at Screening or, in the opinion of the investigator, a hemoglobin level that would make it unsafe for study participation
* Known hypersensitivity to penicillamine
* Female subjects who were nursing, planning a pregnancy, or were known or suspected to be pregnant
* Participants who, in the opinion of the investigator, were not able or willing to comply with study requirements
* Had received a kidney transplant or was currently on dialysis
* Was 6 years of age or older at the time of the Screening visit

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2016-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States
- Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Schwartz GJ, Munoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, Furth SL. New equations to estimate GFR in children with CKD. J Am Soc Nephrol. 2009 Mar;20(3):629-37. doi: 10.1681/ASN.2008030287. Epub 2009 Jan 21. PMID 19158356
- See also: Related Info — http://www.horizonpharma.com/medicines/rare-diseases/procysbi/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety Population: All participants who received at least 1 dose of RP103.
Period: Overall Study
Arm/Group | RP103
Started | 17
Completed | 16
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least 1 dose of RP103.
Arm/Group | RP103
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.80 (5.116)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean White Blood Cell (WBC) Cystine Concentration at Each Visit
Description: Blood samples were taken 30 minutes after the morning RP103 dose at each study visit to determine White Blood Cell (WBC) cystine concentration. WBC cystine concentrations were determined using liquid chromatography.
Time Frame: Day 1, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Month 6, Month 9, Month 12, Month 15, Month 18, Study Exit
Population: Participants <6 years of age who received at least 1 dose of RP103 and who had at least 1 WBC cystine level recorded.
Measure: Mean (Standard Deviation); unit: nmol 1/2 Cystine/mg protein
Arm/Group | RP103
Number analyzed (Participants) | 15
nmol 1/2 Cystine/mg protein
  Day 1 | 3.1709 (2.95209)
  Week 2 | 2.2899 (3.13707)
  Week 4: number analyzed (Participants) | 13
  Week 4 | 1.8474 (1.62820)
  Week 6: number analyzed (Participants) | 13
  Week 6 | 2.3403 (4.31136)
  Week 8: number analyzed (Participants) | 13
  Week 8 | 0.9589 (1.05851)
  Week 10: number analyzed (Participants) | 12
  Week 10 | 1.1219 (1.27413)
  Week 12: number analyzed (Participants) | 13
  Week 12 | 1.1828 (1.31272)
  Month 6: number analyzed (Participants) | 2
  Month 6 | 2.7250 (1.08187)
  Month 9: number analyzed (Participants) | 6
  Month 9 | 2.0196 (1.90931)
  Month 12: number analyzed (Participants) | 13
  Month 12 | 0.8012 (0.59706)
  Month 15: number analyzed (Participants) | 9
  Month 15 | 1.2443 (1.47616)
  Month 18: number analyzed (Participants) | 9
  Month 18 | 0.7356 (0.64027)
  Study Exit: number analyzed (Participants) | 13
  Study Exit | 0.8197 (0.76413)

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Safety was assessed by the incidence of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (SAEs). An AE/adverse experience was any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. For additional information regarding adverse events, please see the safety section of the record.
Time Frame: Day 1 through study exit
Population: Safety population: All participants who received at least 1 dose of RP103.
Measure: Count of Participants; unit: Participants
Arm/Group | RP103
Number analyzed (Participants) | 17
Participants | 17

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Cysteamine
Description: Blood samples were collected and plasma cysteamine concentration was determined using liquid chromatography. The maximum observed plasma concentration (Cmax) of cysteamine was determined directly from the data.
Time Frame: 30 minutes after the morning RP103 dose at Month 6 (prior to Protocol Amendment 1) or 0 (pre-dose), 30 minutes, 2, 3, 4, 6, 8, 10, and 12 hours after the morning RP103 dose at Month 6 for those enrolled under Protocol Amendment 1 or later
Population: Participants age <6 years who received at least 1 dose of RP103 and participated in frequent sampling at the Month 6 visit.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | RP103
Number analyzed (Participants) | 11
mg/L | 1.26 (0.86)

4. Secondary Outcome: Time of the Maximum Observed Plasma Concentration (Tmax) of Cysteamine
Description: Blood samples were collected and plasma cysteamine concentration was determined using liquid chromatography. The time of the maximum observed plasma concentration (Tmax) of cysteamine was determined directly from the data.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | RP103
Number analyzed (Participants) | 11
minutes | 199 (138)

5. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Cysteamine
Description: Blood samples were collected and plasma cysteamine concentration was determined using liquid chromatography. AUC values were estimated using non-compartmental analysis methods. AUClast was defined as the area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (720 minutes). AUCinf was defined as the area under the plasma concentration-versus-time curve from time 0 to infinity.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: min*mg/L
Arm/Group | RP103
Number analyzed (Participants) | 11
min*mg/L
  AUClast | 206 (113)
  AUCinf: number analyzed (Participants) | 10
  AUCinf | 231 (123)

ADVERSE EVENTS:
Time Frame: From Day 1 through study exit
Description: Adverse events (AEs) were defined as any AE with onset following initial drug administration (on Day 1).
Arm/Group | RP103
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 12/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RP103 (N=17)
Gastroenteritis (Infections and infestations) | 5
Catheter Site Infection (Infections and infestations) | 1
Clostridium difficile Colitis (Infections and infestations) | 1
Gastroenteritis Viral (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Electrolyte Imbalance (Metabolism and nutrition disorders) | 2
Failure to Thrive (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Abdominal Distension (Gastrointestinal disorders) | 1
Gastrostomy (Surgical and medical procedures) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Cardiopulmonary Failure (Cardiac disorders) | 1
Fanconi Syndrome (Congenital, familial and genetic disorders) | 1
Hypovolaemic Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RP103 (N=17)
Vomiting (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 6
Breath Odour (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 8
Gastroenteritis (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 3
Catheter Site Infection (Infections and infestations) | 1
Otitis Media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Pyrexia (General disorders) | 4
Granuloma (General disorders) | 1
Medical Device Site Reaction (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Conjunctivitis (Eye disorders) | 1
Strabismus (Eye disorders) | 1
Headache (Nervous system disorders) | 2
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 2
Gastrostomy Closure (Surgical and medical procedures) | 1
Gastrostomy Tube Removal (Surgical and medical procedures) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1
Perineal Erythema (Reproductive system and breast disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights .